CLINICAL TRIAL: NCT02710617
Title: System Accuracy Evaluation of 2 CE-marked Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Other Study IDs: IDT-1542-IU
Record Dates: First submitted 2016-03-11; First posted 2016-03-17 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Device: Blood glucose monitoring systems for point-of-care-testing
  Other Names: Hemocue Glucose 201+ and Hemocue Glucose 201 RT

SUMMARY:
The objective of this study is the evaluation of system accuracy following ISO 15197:2013 (E), clause 6.3 in which accuracy requirements and applicable test procedures for blood glucose monitoring systems intended for self-monitoring of blood glucose by patients are stipulated.

However in this study, system accuracy evaluation will be performed for Hemocue Glucose 201+ and Hemocue Glucose 201 RT which are both glucose monitoring systems for professional use only on behalf of the IDT with one reagent system lot for each BGMS.

Main goal is the evaluation of system accuracy of both of the hemocue Systems. (english)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes or subjects without diabetes
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.
* If blood glucose values < 80 mg/dl or > 300 mg/dl shall be measured after short term alteration in insulin therapy:
* Male or female with type 1 diabetes and intensified insulin therapy or insulin pump therapy.
* Signature of subjects to document consent with these procedures on informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Being unable to give informed consent
* < 18 years
* Legally incompetent
* Being committed to an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent on investigator or sponsor
* If blood glucose values < 80 mg/dl shall be measured after short term alteration in insulin therapy (concentration category 2, see Fehler! Verweisquelle konnte nicht gefunden werden.), subjects with type 1 diabetes, suffering from:
* Coronary heart disease
* Condition after myocardial infarction
* Condition after cerebral events
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
System accuracy criteria (see description) | For each subject, the experimental phase has an expected duration of up to 6 hours
  System accuracy criteria
  * Following ISO 15197:2013 (E), the BGMS shall meet both of the following criteria:
  * Criterion A: 95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 100 mg/dl (5.55 mmol/l) or within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).
  * Each lot shall pass acceptability criterion A.
  * Criterion B: 99 % of individual glucose measured values shall fall within zones A and B of the Consensus Error Grid (CEG) for type 1 diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany